CLINICAL TRIAL: NCT01538966
Title: Comparison of Combination Low-Dose SRL + Daily Pegvisomant Therapy, Low-Dose SRL + Weekly Pegvisomant Therapy, and High-Dose SRL + Weekly Pegvisomant Therapy
Brief Title: Acromegaly Combination Treatment Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Review of the 12-month data showed patients who deviated from protocol with full IRB monitoring and reporting could not be optimally analyzed. Reopening the study for new enrollment is not feasible and the study was terminated with IRB approval.
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Shlomo Melmed, MD, Executive Vice President, Academic Affairs, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro26424; WS2036536 (Other Grant/Funding Number: Pfizer)
Record Dates: First submitted 2012-02-21; First posted 2012-02-27 (Estimated); Results first posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-08

CONDITIONS: Acromegaly
Keywords: acromegaly; pituitary; pegvisomant; somavert; lanreotide; octreotide
MeSH Terms: conditions — Acromegaly; Pituitary Diseases | interventions — pegvisomant; Octreotide; lanreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High dose SRL + weekly Pegvisomant (Active Comparator): High dose of SRL monthly
  * Octreotide LAR 30mg
  * Lanreotide 120mg
  Weekly Pegvisomant (40-120mg/week)
  Interventions: Drug: Pegvisomant; Drug: Octreotide LAR; Drug: Lanreotide
- Low dose SRL + daily Pegvisomant (Active Comparator): Low dose of SRL monthly
  * Octreotide LAR 10mg
  * Lanreotide 60mg
  Daily Pegvisomant (15-60mg/day)
  Interventions: Drug: Pegvisomant; Drug: Octreotide LAR; Drug: Lanreotide
- Low dose SRL + weekly Pegvisomant (Active Comparator): Low dose of SRL monthly
  * Octreotide LAR 10mg
  * Lanreotide 60mg
  Weekly Pegvisomant (40-120mg/week)
  Interventions: Drug: Pegvisomant; Drug: Octreotide LAR; Drug: Lanreotide

INTERVENTIONS:
Drug: Pegvisomant
  Other Names: Somavert
Drug: Octreotide LAR
  Other Names: Sandostatin
Drug: Lanreotide
  Other Names: Somatuline

SUMMARY:
In this study the investigators will evaluate whether combination low dose somatostatin receptor ligand (SRL) and weekly or daily pegvisomant will attain equivalent control of serum insulin-like growth factor (IGF)-1 levels at a lower cost, compared to combination high dose SRL and weekly pegvisomant. Lower doses of therapy will greatly reduce cost of acromegaly therapy.

DETAILED DESCRIPTION:
Subjects will be stratified based on prior response to SRL therapy and then randomized to one of three treatment arms. The study will begin when the combination of octreotide long-acting release (LAR) or lanreotide and pegvisomant is first administered. Study visits will occur every 4 weeks from the start of the study. However, for subjects who cannot make every study visit due to distance, the study team will facilitate monthly blood draws at their local Quest laboratory facility.

After the 24 weeks of combination therapy, subjects with a controlled IGF-1 will then start pegvisomant monotherapy at the same dose and schedule that they attained normalization in combination therapy. IGF-1 levels, liver function test, and blood glucose will be performed monthly. Magnetic resonance imaging (MRI) will be performed at the conclusion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with acromegaly who have not had surgery or medical therapy
* Acromegaly patients who are at least 3 months post surgery, who are/are not receiving adjuvant medical therapy
* Acromegaly patients on SRL monotherapy with normal or elevated IGF-1 levels
* Acromegaly patients on Pegvisomant monotherapy with normal or elevated IGF-1 levels.
* Acromegaly patients who have received SRL and dopamine agonist therapy, after a 6 week washout period of the dopamine agonist.
* Acromegaly patients on combination therapy with maximum doses of SRL and Pegvisomant (daily or weekly
* Normal liver function tests before randomization to treatment
* The patient has had appropriate dynamic testing of the pituitary axis and, if applicable, is receiving appropriate hormone replacement therapy.

Exclusion Criteria:

* The patient harbors a macroadenoma with visual field defects due to chiasmatic compression
* The patient has clinically significant hepatic abnormalities and/or aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) above 3 times the upper limit of normal at the baseline visit.
* The patient had pituitary surgery within 3 months prior to study entry
* The patient had radiotherapy within 12 months prior to study entry
* The patient has abnormal CBC and chemistry panel at the baseline visit, any other medical condition(s) or laboratory findings that, in the opinion of the investigator, might jeopardize the patient's safety.
* The patient has a known hypersensitivity to any of the test materials or related compounds.
* The patient has a history of, or known current problems with alcohol or drug abuse.
* The patient has any mental condition rendering the patient unable to understand the nature, scope, and possible consequences of the study, and/or evidence of an uncooperative attitude.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2012-03-29 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shlomo Melmed, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Result] Bonert V, Mirocha J, Carmichael J, Yuen KCJ, Araki T, Melmed S. Cost-Effectiveness and Efficacy of a Novel Combination Regimen in Acromegaly: A Prospective, Randomized Trial. J Clin Endocrinol Metab. 2020 Sep 1;105(9):dgaa444. doi: 10.1210/clinem/dgaa444. PMID 32754748

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Dose SRL + Weekly Pegvisomant | Low Dose SRL + Daily Pegvisomant | Low Dose SRL + Weekly Pegvisomant
Started | 23 | 26 | 27
Completed | 15 | 14 | 23
Not Completed | 8 | 12 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose SRL + Weekly Pegvisomant | Low Dose SRL + Daily Pegvisomant | Low Dose SRL + Weekly Pegvisomant | Total
Number analyzed (Participants) | 15 | 14 | 23 | 52
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.6 (17.6) | 52.9 (12.1) | 48.0 (13.3) | 49.5 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 14 | 32
  Male | 5 | 6 | 9 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 1 | 0 | 0 | 1
  White | 14 | 13 | 18 | 45
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cost Effectiveness
Description: We evaluated cost-effectiveness of combination low-dose SRL and weekly or daily pegvisomant compared to combination high-dose SRL and weekly pegvisomant by assessing cost of therapy per month in each treatment arm among patients who achieved normal IGF-1 levels.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: US dollars/month
Arm/Group | High Dose SRL + Weekly Pegvisomant | Low Dose SRL + Daily Pegvisomant | Low Dose SRL + Weekly Pegvisomant
Number analyzed (Participants) | 15 | 14 | 23
US dollars/month | 14,261.33 (1,645.49) | 22,542.86 (11,158.49) | 9,836.52 (1,374.99)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events were recorded during weekly phone calls with study staff and confirmed at each monthly study visit in person or on the phone.
Arm/Group | High Dose SRL + Weekly Pegvisomant | Low Dose SRL + Daily Pegvisomant | Low Dose SRL + Weekly Pegvisomant
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 1/23
Other Adverse Events (participants affected / at risk) | 4/15 | 2/14 | 9/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose SRL + Weekly Pegvisomant (N=15) | Low Dose SRL + Daily Pegvisomant (N=14) | Low Dose SRL + Weekly Pegvisomant (N=23)
Tuberculosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose SRL + Weekly Pegvisomant (N=15) | Low Dose SRL + Daily Pegvisomant (N=14) | Low Dose SRL + Weekly Pegvisomant (N=23)
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 6
Headache (Nervous system disorders) | 4 | 0 | 2
Joint pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 4
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Swelling (General disorders) | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/66/NCT01538966/Prot_SAP_000.pdf